CLINICAL TRIAL: NCT02840994
Title: A Phase 1 Trial of CV301 in Combination With Anti- PD-1 Therapy in Subjects With Non-Small Cell Lung Cancer
Brief Title: A Trial of CV301 in Combination With Anti-PD-1 Therapy in Subjects With Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CV301-2015-201; MAGNI-LUNG-01 (Other: Bavarian Nordic, Inc.)
Record Dates: First submitted 2016-07-18; First posted 2016-07-21 (Estimated); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
Keywords: CV301, NSCLC, Pembrolizumab, Nivolumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CV301 + Pembrolizumab (Experimental): CV301 + Pembrolizumab (Phase 1b portion of the trial)
  Interventions: Biological: CV301; Biological: Pembrolizumab
- CV301 + Nivolumab (Experimental): CV301 + Nivolumab (Phase 1b portion of the trial)
  Interventions: Biological: CV301; Biological: Nivolumab

INTERVENTIONS:
Biological: CV301
Biological: Pembrolizumab
  Other Names: KEYTRUDA
  Arms: CV301 + Pembrolizumab
Biological: Nivolumab
  Other Names: OPDIVO
  Arms: CV301 + Nivolumab

SUMMARY:
The objective of the proposed clinical trial is to investigate the safety and tolerability of CV301 in combination with Anti-PD1-Therapy in subjects with non-small cell lung cancer (NSCLC).

The clinical trial is designed to evaluate the possible enhanced antitumor activity of CV301 with Anti-PD1-Therapy. The rationale for combining CV301 with Anti-PD1-Therapy is based on the hypothesis that CV301 can induce specific immune response in the tumor, and that in combination, Anti-PD1-Therapy may augment the T cell-mediated immune response generated by CV301 by blocking the inhibitory signal of the PD-1.

The trial will include a Phase 1 portion and a Phase 1b portion with 2 cohorts. The Phase 1 portion is a dose escalation part to assess the safety and tolerability of CV301 alone, prior to moving into the combination with Anti-PD1-Therapy (the Phase 1b component).

The following Phase 1b portion of the trial aims to test the safety and tolerability of the combination treatment using a two cohort approach with cohort 1 receiving CV301 plus Nivolumab and cohort 2 receiving CV301 plus Pembrolizumab.

ELIGIBILITY:
Inclusion criteria for the Phase 1:

1. Subjects must have a metastatic or unresectable locally advanced malignant solid tumor, histologically confirmed by the Laboratory of Pathology, NCI. Efforts will be made, as much as possible, to enroll subjects with tumor types with known increased expression of CEA or MUC-1 (such as lung, breast, ovarian, prostate, colorectal, pancreatic, bladder, gastric, cervix, etc.).
2. Subjects may have measurable or nonmeasurable but evaluable disease. Subjects with surgically resected or ablated metastatic disease at high risk of relapse are also eligible.

   Prior therapy: Subjects must have completed or had disease progression on at least one prior line of disease-appropriate therapy for locally advanced or metastatic disease, or not be candidates for therapy of proven efficacy for their disease.
3. Subjects with EGFR or ALK genomic tumor aberrations should have disease progression on FDA-approved therapy for these aberrations.
4. There should be a minimum of 4 weeks from any prior chemotherapy, immunotherapy and/or radiation, with the exception of hormonal therapy for prostate and breast cancers, HER2-directed therapy for HER2+ breast cancer (3+ IHC or FISH+), maintenance therapy for colorectal or pancreatic cancer, and erlotinib therapy in EGFR-mutated lung cancer under the condition that subjects are on these therapies for at least two months before start of trial treatment. There should be a minimum of 6 weeks from any prior antibody therapies (such as ipilimumab or Anti-PD1/PDL1) due to prolonged half-life.
5. Subjects must have recovered (Grade 1 or baseline) from any clinically significant toxicity associated with prior therapy. Typically, this is 3-4 weeks for subjects who most recently received cytotoxic therapy, except for nitrosoureas and mitomycin C, for which 6 weeks is needed for recovery.
6. Men or women, age ≥ 18 years.
7. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1 or Karnofsky ≥ 70%, (see Section 19.1, Appendix I and Section 19.2, Appendix II).
8. Subjects must have normal organ and marrow function as defined below

   a. Serum creatinine ≤ 1.5 x upper limit of normal (ULN) OR creatinine clearance (CrCl) ≥ 40 mL/min (if using the Cockcroft-Gault formula below): i. Female CrCl = [(140 - age in years) x weight in kg x 0.85] / [72 x serum creatinine in mg/dL] ii. Male CrCl = [(140 - age in years) x weight in kg x 1.00] / [72 x serum creatinine in mg/dL] b. Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) ≤ 3 x the ULN c. Total bilirubin ≤ 1.5 x ULN OR in subjects with Gilbert's syndrome, a total bilirubin ≤ 3.0 x ULN d. Hematological eligibility parameters (within 16 days of starting therapy): i. Platelet count ≥ 100,000/µL ii. Absolute neutrophil count (ANC) ≥ 1/ µL
9. Subjects must have baseline pulse oximetry > 90% on room air.
10. The effects of CV301 on the developing human fetus are unknown. For this reason, women of child-bearing potential (WOCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to trial entry and for the duration of trial participation and for a period of 4 months after the last vaccination. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this trial, she should inform her treating physician immediately.
11. Subjects with prostate cancer must continue to receive GnRH agonist therapy (unless orchiectomy has been done).
12. Subjects must be able to understand and be willing to sign a written informed consent document.

Inclusion criteria for the Phase 1b:

1. Histologically confirmed non-squamous NSCLC, metastatic or unresectable locally advanced. Actionable EGFR mutations and ALK/ROS-1 translocations targetable with FDA approved therapy must be evaluated and found not to be present by standard methods. Expression of PD-L1 must have been determined with a validated method or tumor sample must be available for PD-L1 expression determination.
2. Patient population:

   • Phase 1b, Cohort 1 (Nivolumab + CV301): Patients with progression on or after prior platinum, with or without switch maintenance chemotherapy are eligible

   • Phase 1b, Cohort 2 (Pembrolizumab + CV301): Patients must have been on Pembrolizumab as first-line therapy for NSCLC as per FDA approved indications in first line for at least 11 weeks and assessed by RECIST to have CR, PR, or SD at week 12 (+/- 1 week).

   As of June 2017, FDA-approved indications for front-line treatment include 2 indications for Pembrolizumab:
   * As a single agent for the first-line treatment of patients with metastatic NSCLC whose tumors have high PD-L1 expression (Tumor Proportion Score (TPS) ≥50%) as determined by an FDA-approved test, with no EGFR or ALK genomic tumor aberrations.
   * In combination with pemetrexed and carboplatin, as first-line treatment of patients with metastatic nonsquamous NSCLC. This indication is approved under accelerated approval based on tumor response rate and progression-free survival. Continued approval for this indication may be contingent upon verification and description of clinical benefit in the confirmatory trials.

   Pemetrexed single agent maintenance after the initial 4 cycles of pemetrexed in combination with carboplatinum and Pembrolizumab is allowed and optional as per investigator or institutional standard practice.
3. In case of metastatic recurrence of a previous early stage NSCLC, any chemotherapy or radiation therapy must have finalized more than 12 months before the start of the first-line treatment, either Pembrolizumab alone or in combination with pemetrexed and carboplatinum.
4. ECOG performance status 0 and 1.
5. Men or women, age ≥ 18 years
6. Have normal organ and marrow function as defined below:

   * Serum creatinine ≤ 1.5 x upper limit of normal (ULN) OR creatinine clearance (CrCl) ≥ 40 mL/min (if using the Cockcroft-Gault formula below):

     i. Female CrCl = [(140 - age in years) x weight in kg x 0.85] / [72 x serum creatinine in mg/dL] ii. Male CrCl = [(140 - age in years) x weight in kg x 1.00] / [72 x serum creatinine in mg/dL]
   * ANC > 1/µL
   * Platelets ≥ 100 000/µL
   * Hemoglobin > 9 g/dL
   * Total bilirubin ≤ 1.5 x institutional ULN or direct bilirubin < ULN if total bilirubin > 1.5-3.0 x ULN
   * AST/ALT < 2.5 × institutional ULN, or < 5 x ULN, if liver metastases are present
7. Have measurable disease by computed tomography (CT)/Magnetic resonance imaging (MRI) per RECIST 1.1.
8. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures.
9. Able to understand and be willing to sign a written informed consent document.
10. WOCBP must use appropriate method(s) of contraception. WOCBP should use an adequate method to avoid pregnancy for 23 weeks (30 days plus the time required for Nivolumab to undergo five half-lives) after the last dose of investigational drug (Phase 1b, Cohort 1). WOCBP should use an adequate method to avoid pregnancy for at least 4 months (as per approved Pembrolizumab prescribing information) after the last dose of investigational drug (Phase 1b, Cohort 2).
11. Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of β-human choriogonadotropin (HCG)) at screening. They must have confirmation by a negative urine pregnancy test within 24 hours prior to the first dose of Nivolumab (Phase 1b, Cohort 1), or within 24 hours prior to the first dose of Pembrolizumab (Phase 1b, Cohort 2) in the setting of this trial.
12. Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. Men receiving Nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 31 weeks after the last dose of investigational product. Women who are not of childbearing potential (ie, who are postmenopausal or surgically sterile) as well as azoospermic men, do not require contraception.
13. Subjects must have, prior to trial treatment, at least 10 unstained tissue slides (or a tissue block from which 10 slides can be cut) from a prior biopsy or surgical resection for submission for research purposes.

Optional for Phase 1b.

Exclusion Criteria for all Phases:

1. Subjects with EGFR mutations, ALK or ROS-1 translocations candidates to targeted therapy.
2. Squamous histology of NSCLC.
3. Other concurrent investigational agents (subjects are eligible to enroll 4 weeks after completion of prior investigational agent).
4. More than 1 prior chemotherapy regimen for locally advanced or metastatic NSCLC with the exception of the Phase 1 portion, in which multiple therapies are allowed in all tumor types. Any prior chemotherapy regimen different from pemetrexed-carboplatinum in combination with Pembrolizumab as first-line chemotherapy for candidates to Pembrolizumab maintenance of first line (Phase 1b).
5. Concurrent chemotherapy or radiotherapy or other immunotherapy not explicitly allowed by inclusion criteria for that phase of trial.
6. Subjects treated with PD-1/L1 or any other experimental immunotherapeutic agents outside the parameters established in the inclusion criteria, are excluded from enrollment into Phase 1b, but can be enrolled into Phase 1.
7. Other malignancy within last 5 years with an estimated risk of recurrence higher than 50%. Examples of low risk of recurrence malignancies are non-melanoma skin cancer, in situ cervical, superficial bladder cancer, colorectal cancer stage I and II, breast cancer stages I and II, prostate cancer stages I and II, etc.
8. Patients with metastatic lesions in the brain.
9. History of allergy or untoward reaction to prior vaccination with vaccinia virus, aminoglycoside antibiotics or egg products; history of allergy to smallpox vaccination.
10. Active infection within 72 hours prior to vaccination.
11. Subjects should have no known evidence of being immunocompromised as listed below:

    1. Human immunodeficiency virus (HIV) positivity, chronic hepatitis infection, including hepatitis B and C virus
    2. Active, known or suspected autoimmune disease. Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger
    3. Immunosuppressive therapy post-organ transplant
    4. Asplenia is an exclusion for Phase 1b, but is not an exclusion for Phase 1.
12. Altered immune function, including, but not limited to: inflammatory bowel disease; active infectious enteritis; eosinophilic enteritis; lupus erythematosus; ankylosing spondylitis; scleroderma; multiple sclerosis. These criteria do not include all diseases with an immune-related component, but are not auto-immune in nature or have a primary alteration in the general immune function that may interfere with the vaccine mechanism of action, for example celiac disease.
13. Concurrent chronic use of systemic steroids, except for physiologic doses of systemic steroids for replacement, defined as 5 mg of prednisone per day or equivalent, or local (topical, nasal, ophthalmic or inhaled) steroid use or prior concomitant use with chemotherapy. Systemic steroids must have been discontinued ≥ 2 weeks prior to first treatment. Prior use of corticoids in short-term schemes (duration shorter than 3 days) for indications such as prophylaxis of reactions to intravenous contrast for imaging studies or chemotherapy-related AEs are not considered part of this exclusion. Prior use of corticoids for brain metastasis ending before day -14 is not considered part of this exclusion criteria.
14. Subjects with interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity.
15. Pregnant or breastfeeding women.
16. Clinically significant cardiomyopathy, coronary disease, heart failure New York Heart Association class III or IV, or cerebrovascular accident within 1 year.
17. Uncontrolled intercurrent illness, which would interfere with the ability of the subject to carry out the treatment program.
18. Any other condition, which would, in the opinion of the Principal Investigator or Medical Monitor, indicate the subject is a poor candidate for treatment with CV301 or would jeopardize the subject or the integrity of the data obtained.
19. Medical or psychological impediment to compliance with protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of CV301 alone and in combination determined by incidence of dose-limiting toxicities (DLTs) | Through study completion, up to 2 years
  Safety and tolerability following administration of CV301 alone (Phase 1) and in combination with Nivolumab or Pembrolizumab (Phase 1b), respectively, as determined by the incidence of dose-limiting toxicities (DLTs).

CONTACTS AND LOCATIONS:
Overall Officials: Cesar Pico-Navarro, MD, Study Director — Bavarian Nordic
Locations (7):
- United States (7):
  - H. Lee Moffitt Cancer Center & Research Institute, Inc., Tampa, Florida
  - Investigative Clinical Research of Indiana, Indianapolis, Indiana
  - Metairie Oncologist, LLC, Metairie, Louisiana
  - NCI, Bethesda, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Novant Health Oncology Specialists, Winston-Salem, North Carolina
  - Millennium Oncology, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Derived] Rajan A, Gray JE, Devarakonda S, Birhiray R, Korchin B, Menius E, Donahue RN, Schlom J, Gulley JL. Phase 1 trial of CV301 in combination with anti-PD-1 therapy in nonsquamous non-small cell lung cancer. Int J Cancer. 2023 Feb 1;152(3):447-457. doi: 10.1002/ijc.34267. Epub 2022 Sep 9. PMID 36054490